CLINICAL TRIAL: NCT01389505
Title: Structural and Functional Evaluation of the Macula in Patients With Proliferative Diabetic Retinopathy Treated With Panretinal Photocoagulation and Bevacizumab (Avastin ®)
Brief Title: Bevacizumab as Adjunctive Treatment to Laser Panretinal Photocoagulation for Proliferative Diabetic Retinopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Coracao (Other Government)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: University of Sao Paulo, Faculdade de Medicina da Universidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CONEP16249; CONEP16249 (Other: CONEP16249)
Record Dates: First submitted 2011-07-05; First posted 2011-07-08 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-01

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Proliferative Diabetic Retinopathy; Bevacizumab; Panretinal Photocoagulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panretinal photocoagulation (Active Comparator): Group 1: Panretinal photocoagulation treatment (PRP) at month-0 that can be repeated after month-3.
  Interventions: Procedure: Panretinal photocoagulation
- Bevacizumab + Panretinal Photocoagulation (PRP) (Experimental): Group 2: Bevacizumab intravitreous injections plus PRP
  Interventions: Procedure: Procedure: Panretinal Photocoagulation (PRP) Drug: Intravitreous injection of Bevacizumab

INTERVENTIONS:
Procedure: Panretinal photocoagulation — Three episodes of panretinal photocoagulation with one week of interval
  Arms: Panretinal photocoagulation
Procedure: Procedure: Panretinal Photocoagulation (PRP) Drug: Intravitreous injection of Bevacizumab — Intravitreous injection of Bevacizumab 1 week before and the other at the same day of the third episode of PRP
  Arms: Bevacizumab + Panretinal Photocoagulation (PRP)

SUMMARY:
This is a prospective, randomized and comparative study is to quantify the functional and structural alterations of the macula in patients with proliferative Diabetic Retinopathy submitted to laser photocoagulation and to evaluate the efficacy of intravitreal bevacizumab as a adjuvant therapy in preventing the adverse events of that procedure. The patients with proliferative Diabetic Retinopathy (DR) with indication of binocular laser photocoagulation will be examined by ophthalmologists who will measure the visual acuity and contrast sensitivity, perform slit lamp examination, fundus examination and optic coherence tomography before and after laser photocoagulation. Laser photocoagulation will be performed in both eyes according Early Treatment Diabetic Retinopathy Study that advocate the realization of 3 episodes of laser photocoagulation in 3 weeks. This comparative study analyses the effect of intravitreal bevacizumab one week before laser photocoagulation and one, three and six months after the randomization visit. The fellow eye will be submitted only to laser photocoagulation and will be considered as control. It is estimated a sample of 30 patients. All procedures, purposes and methods will be explained to all patients.

DETAILED DESCRIPTION:
The current gold standard for the treatment of proliferative diabetic retinopathy is panretinal photocoagulation. Therefore this study is designed using both treatments in the same patient: intravitreal Bevacizumab plus panretinal photocoagulation in one eye, compared to panretinal photocoagulation alone in the contralateral eye. These patients had their visual acuity and contrast vision measured and complete ophthalmological examination was performed, including macular slit lamp examination, fluorescein angiography and optical coherence tomography.

Patients with similar proliferative diabetic retinopathy without high risk characteristics receive laser therapy in both eyes and intravitreal Bevacizumab injections in one eye. For the Bevacizumab injections, numbing drops, antibiotic drops, and drops to dilate the pupil, and possibly and anesthetic injection, are put in the eye before the medicine is injected into the vitreous. Patients return for follow-up visits 1 day, 1 and 4 weeks after the injection, and then 3 and 6 months. Patients whose condition does not improve may undergo new evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Proliferative diabetic retinopathy eyes.
* Best Corrected-Visual Acuity at baseline > 20/320 in the study eye.
* Patients with and without diabetic macular edema
* Type II diabetic subjects as defined by the World Health Organization
* aged ≥ 18 years.
* Women must be using effective contraception
* Ability to provide written informed consent.
* Indication of panretinal photocoagulation in both eyes

Exclusion Criteria:

* Vitreous hemorrhage or pre-retinal hemorrhage
* Eyes with prior scatter (panretinal) or focal/grid photocoagulation, within the previous 6 months.
* Atrophy/scarring/fibrosis/ hard exudates involving the center of the macula.
* Cataract
* Any intraocular surgery within 6 months before trial enrollment.
* Previous vitrectomy.

Any of the following underlying systemic diseases:

History or evidence of severe cardiac disease or previous thrombus-embolic event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Functional Macular Evaluation | 24 weeks
  During this 24 weeks of follow-up the Visual acuity (ETDRS), Contrast vision will be measured at baseline, 4, 12 and finally at 24 week

SECONDARY OUTCOMES:
Structural Macular Evaluation | 24 weeks
  During the 24 weeks of follow-up the following measured will be made: Optical coherence tomography, need of vitrectomy, need panretianal photocoagulation retreatment, adverse events, recurrence of neovascularizaton, need or additional focal and grid macular laser for diabetic macular edema

CONTACTS AND LOCATIONS:
Overall Officials: Walter Y Takahashi, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Preti RC, Mutti A, Ferraz DA, Zacharias LC, Nakashima Y, Takahashi WY, Monteiro ML. The effect of laser pan-retinal photocoagulation with or without intravitreal bevacizumab injections on the OCT-measured macular choroidal thickness of eyes with proliferative diabetic retinopathy. Clinics (Sao Paulo). 2017 Feb 1;72(2):81-86. doi: 10.6061/clinics/2017(02)03. PMID 28273240
- [Derived] Preti RC, Ramirez LM, Monteiro ML, Carra MK, Pelayes DE, Takahashi WY. Contrast sensitivity evaluation in high risk proliferative diabetic retinopathy treated with panretinal photocoagulation associated or not with intravitreal bevacizumab injections: a randomised clinical trial. Br J Ophthalmol. 2013 Jul;97(7):885-9. doi: 10.1136/bjophthalmol-2012-302675. Epub 2013 May 17. PMID 23686001